CLINICAL TRIAL: NCT05684549
Title: Effects of Coronavirus Infection (COVID-19) on the Timing and Prognosis of Radical Surgery in Patients With Early-stage Lung Cancer
Brief Title: Coronavirus Infection (COVID-19) and Radical Surgery in Patients With Early-stage Lung Cancer
Acronym: COVIDLungSurg
Status: Active, not recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Professor, Ruijin Hospital
Other Study IDs: RTS-017
Record Dates: First submitted 2023-01-12; First posted 2023-01-13 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Surgery; Corona Virus Infection
Keywords: Lung cancer; Surgery; Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stage I/II lung cancer patients: Patients with stage I/II lung cancer will receive radical surgery.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study, no intervention

SUMMARY:
The goal of this observational study is to learn about the effects of coronavirus infection in patients with early-stage lung cancer. The main question it aims to answer is whether the interval of surgery and COVID-19 infection will affect the surgery and prognosis of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed stage I and stage II lung cancer, who are about to receive wedge resection, segmental resection, sleeve resection, lobectomy, or pneumonectomy under general anaesthesia.
* Volunteer to participate in the study with good compliance. Able to complete the observation and follow-up and have signed the informed consent.
* ASA score: I-III;
* Cardiopulmonary functions meet the requirements of radical operation for lung cancer with normal liver and kidney functions.

Exclusion Criteria:

* Neurologic, mental illness or mental disorder which is hard to control, poor compliance, unable to cooperate or describe the treatment response;
* Clinically diagnosed stage III and stage IV lung cancer or patients who received neoadjuvant treatment before surgery;
* Patients developed symptoms alike coronavirus infection but are not confirmed by viral RNA detection by quantitative RT-PCR or antigen testing kits.
* Serious heart, lung, liver and kidney dysfunction and unable to tolerate the operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically diagnosed stage I or stage II lung cancer who are about to receive radical surgery.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative morbidity | postoperative in-hospital stay up to 30 days
  rate of perioperative complications, mainly include: pneumonia, respiratory failure, pulmonary embolism, arrhythmia, sepsis, cerebrovascular accident, myocardial injury, acute kidney injury.

SECONDARY OUTCOMES:
postoperative hospital stay | postoperative in-hospital stay up to 30 days
  length of postoperative hospitalization
operation time | At operation day
  duration of operation
R0 rate | postoperative in-hospital stay up to 30 days
  R0 resection rate
blood loss | At operation day
  blood loss in the operation
30-day mortality | postoperative in-hospital stay up to 30 days
  30-day mortality after surgery
quality of life | postoperative in-hospital stay up to 30 days
  postoperative quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Niu Z, Zhu F, Cao Y, Luo C, Liu D, Wang C, Qiu Z, Peng L, Du M, Jin R, Yan Y, Dong D, Jing H, Wang X, Guo W, Guo Z, Li C, Han D, Zhang Y, Xiang J, Du H, Chen K, Yin Z, Yang J, Zhong W, Zhou Y, Wang M, Ma D, Li H. Impact of coronavirus disease 2019 on surgery in patients with early-stage lung cancer: the COVIDLungSurg prospective cohort study. Transl Lung Cancer Res. 2025 May 30;14(5):1677-1687. doi: 10.21037/tlcr-2024-1276. Epub 2025 May 28. PMID 40535078